CLINICAL TRIAL: NCT05279508
Title: Make My Day: an eHealth Supported Stroke Prevention Program for Primary Health Care Preventing Stroke and Supporting Everyday Activities
Brief Title: Make My Day - a Stroke Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ann-Helen Patomella, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KI2020-00175
Record Dates: First submitted 2022-01-26; First posted 2022-03-15 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Non-communicable Disease
Keywords: Primary prevention; Engaging everyday activities; Occupational therapy; Primary healthcare
MeSH Terms: conditions — Stroke; Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and assessor are blinded to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention treatment group (Experimental): 10 week stroke prevention program with six group sessions on pre-set themes targeting modifiable stroke risk factors . The group sessions are chaired by health professionals but also consists of peer learning to support change in lifestyle habits and activity patterns and reduce stroke risk. The change process is supported with a mHealth application for daily registrering of six domains; stroke risk factors, EEA, stress and goal achievement.
  A lifestyle and stroke risk analysis will be performed at baseline measures, at follow up and at 12 month follow up.
  Interventions: Behavioral: Make My Day - stroke prevention program
- Standard treatment group (No Intervention): Usual care within primary healthcare. At baseline, follow up and at 12 month follow up a lifestyle and stroke risk analysis will be conducted.

INTERVENTIONS:
Behavioral: Make My Day - stroke prevention program — A stroke prevention program within primary healthcare
  Arms: Prevention treatment group

SUMMARY:
The purpose of this study is to evaluate the effects of a person-centered stroke prevention program implemented in primary healthcare. It is a primary prevention program aiming to reduce stroke risk and thereby prevent stroke through the enabling of lifestyle changes by introducing health beneficial engaging everyday activities promoting healthy activities and habits.

DETAILED DESCRIPTION:
This study is a single-blind randomized control trial with the aim to evaluate the effects of a stroke prevention program, Make My Day (MMD), in comparison to ordinary primary healthcare services for people at risk for stroke. The MMD prevention program aims to reduce modifiable stroke risk factors and the future risk of stroke by introducing health beneficial engaging everyday activities enabling lifestyle changes and promoting healthy activity patterns and habits. It also includes a mHealth application consisting of six domains for registering daily activities, experiences and behaviours: Goal achievements, Physical activity, Engaging everyday activities, Tobacco and alcohol use, Stress levels and Dietary habits, to increase health literacy and awareness of current habits and to foster self-management.

Engaging everyday activities (EEA´s) are activities the person perceives as valuable, meaningful, and purposeful, as well as provide positive feelings and a sense of participation. EEA´s are performed regularly and are a part of a person's life and depending on the activity it may or may not contribute to health.

The MMD prevention program is person-centered group interventio with health professionals as interventionists. The program starts with an individual meeting at baseline with a lifestyle analysis that includes formulating individual activity goals. Follow-up assessment is done one week after the last group session. There are 6 group sessions where each session has a pre-set theme e.g. stroke risk, engaging everyday activities, physical activity, diet, life habits and routines. Five group-sessions will be conducted over a five week period with a booster session after another five weeks, in total 10 weeks.

The MMD prevention program is a theoretically grounded, complex intervention developed in accordance with the Medical Research Council (MRC) guidelines for developing complex interventions. And in line with the MRC guidelines a feasibility and pilot study have already been conducted. To enable reduction of stroke risk and achieve healthy lifestyle habits the MMD program uses strategies based on behavioural change theories. Behaviour change derives from the interaction process between the person, the environment, and the action. Key in the MMD-program is the incorporation of health beneficial EEA´s, either to incorporate new health beneficial EEA´s or to alter current non health beneficial EEA´s.

ELIGIBILITY:
Inclusion Criteria:

* Three or more high stroke risk factors on the Stroke Risk scorecard
* Motivated for lifestyle change
* Motivated for participating in a digital lifestyle prevention (including user of a smartphone or tablet)
* Between 55-75 years of age and without a diagnosis of dementia or cognitive impairment hindering participation

Exclusion Criteria:

* Previously stroke or TIA
* Lack of understanding the Swedish language

Other:

* All participants may choose to interrupt their participation in the study at any time.
* The researcher can also discontinue a participant's participation based on health issues or reasons that might jeopardize that person's safety. Reasons for interruption will be recorded.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-04-09 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Risk for stroke | At baseline
  Risk for stroke is measured with the Swedish version of the Stroke riskometer. The Stroke riskometer uses an algoritm to estimate the 5-year and 10-year stroke risk from multiple choice questions on lifestyle habits and medical history. The result is given in % for both 5-year and 10-year and higher % means higher risk.
Risk for stroke | at 10week follow up
  Risk for stroke is measured with the Swedish version of the Stroke riskometer. The Stroke riskometer uses an algoritm to estimate the 5-year and 10-year stroke risk from multiple choice questions on lifestyle habits and medical history. The result is given in % for both 5-year and 10-year and higher % means higher risk.
Risk for stroke | At 12-month follow up
  Risk for stroke is measured with the Swedish version of the Stroke riskometer. The Stroke riskometer uses an algoritm to estimate the 5-year and 10-year stroke risk from multiple choice questions on lifestyle habits and medical history. The result is given in % for both 5-year and 10-year and higher % means higher risk.

SECONDARY OUTCOMES:
Participation in engaging everyday activities | At baseline
  Participation in engaging everyday activities measured with Canadian Occupational Performance Measure (COPM). Five activities are listed and performance and satisfaction are scored between 1-10. 1 means either not able to perform or not satisfied at all and 10 means either performs extremely well or extremely satisfied.
Participation in engaging everyday activities | At 10-week follow up
  Participation in engaging everyday activities measured with Canadian Occupational Performance Measure (COPM). Five activities are listed and performance and satisfaction are scored between 1-10. 1 means either not able to perform or not satisfied at all and 10 means either performs extremely well or extremely satisfied.
Participation in engaging everyday activities | At 12-month follow up
  Participation in engaging everyday activities measured with Canadian Occupational Performance Measure (COPM). Five activities are listed and performance and satisfaction are scored between 1-10. 1 means either not able to perform or not satisfied at all and 10 means either performs extremely well or extremely satisfied.
Self rated life satisfaction | At baseline
  Self rated life satisfaction measured with LiSat-11. A questionnaire with 11 questions with a scale 1-6.
  1 means unsatisfied and 6 means very satisfied
Self rated life satisfaction | At 10-week follow up
  Self rated life satisfaction measured with LiSat-11. A questionnaire with 11 questions with a scale 1-6.
  1 means unsatisfied and 6 means very satisfied
Self rated life satisfaction | At 12-month follow up
  Self rated life satisfaction measured with LiSat-11. A questionnaire with 11 questions with a scale 1-6.
  1 means unsatisfied and 6 means very satisfied
Self rated health | At baseline
  Self rated health measured with EQ-5D. A questionnaire on self rated health with question on 5 health defining domain with a scale 1-3. 1 means no problems and 3 means extreme problems. Also an analog scale (VAS) ranging 0-100. 100 means best possible health and 0 means worst possible health.
  1 means unsatisfied and 6 means very satisfied
Self rated health | At 10-week follow up
  Self rated health measured with EQ-5D. A questionnaire on self rated health with question on 5 health defining domain with a scale 1-3. 1 means no problems and 3 means extreme problems. Also an analog scale (VAS) ranging 0-100. 100 means best possible health and 0 means worst possible health.
  1 means unsatisfied and 6 means very satisfied
Self rated health | At 12-month follow up
  Self rated health measured with EQ-5D. A questionnaire on self rated health with question on 5 health defining domain with a scale 1-3. 1 means no problems and 3 means extreme problems. Also an analog scale (VAS) ranging 0-100. 100 means best possible health and 0 means worst possible health.
  1 means unsatisfied and 6 means very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Helen Patomella, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholms Sjukhem, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malstam E, Asaba E, Akesson E, Guidetti S, Patomella AH. 'Weaving lifestyle habits': Complex pathways to health for persons at risk for stroke. Scand J Occup Ther. 2022 Feb;29(2):152-164. doi: 10.1080/11038128.2021.1903991. Epub 2021 Apr 4. PMID 33813996
- [Background] Patomella AH, Guidetti S, Malstam E, Eriksson C, Bergstrom A, Akesson E, Kottorp A, Asaba E. Primary prevention of stroke: randomised controlled pilot trial protocol on engaging everyday activities promoting health. BMJ Open. 2019 Nov 2;9(11):e031984. doi: 10.1136/bmjopen-2019-031984. PMID 31678952
- [Background] Patomella AH, Farias L, Eriksson C, Guidetti S, Asaba E. Engagement in Everyday Activities for Prevention of Stroke: Feasibility of an mHealth-Supported Program for People with TIA. Healthcare (Basel). 2021 Jul 30;9(8):968. doi: 10.3390/healthcare9080968. PMID 34442105
- [Background] Asaba E, Bergstrom A, Patomella AH, Guidetti S. Engaging occupations among persons at risk for stroke: A health paradox. Scand J Occup Ther. 2022 Feb;29(2):116-125. doi: 10.1080/11038128.2020.1829036. Epub 2020 Oct 6. PMID 33021851
- [Background] Patomella AH, Guidetti S, Hagstromer M, Olsson CB, Jakobsson E, Nilsson GH, Akesson E, Asaba E. Make My Day: primary prevention of stroke using engaging everyday activities as a mediator of sustainable health - a randomised controlled trial and process evaluation protocol. BMJ Open. 2023 Dec 6;13(12):e072037. doi: 10.1136/bmjopen-2023-072037. PMID 38056945
- [Derived] Johnsson C, Asaba E, Guidetti S, Akesson E, Hagstromer M, Patomella AH. Make My Day - Stroke Prevention Grounded in Engaging Everyday Activities in Primary Healthcare - A Single-Blinded Randomised Controlled Trial. J Prim Care Community Health. 2025 Jan-Dec;16:21501319251385889. doi: 10.1177/21501319251385889. Epub 2025 Nov 2. PMID 41178128